CLINICAL TRIAL: NCT02146742
Title: A Double Blind, Randomized and Placebo Controlled Ascending Single Oral Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of ASP1707 in Healthy Young Japanese Male Subjects
Brief Title: A Study to Assess the Effects of Single Ascending Doses of ASP1707 in Healthy Young Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1707-CL-0002; 2010-024040-15 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Healthy Subjects
Keywords: ASP1707; Japanese subjects; Safety; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — opigolix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. ASP1707 lowest dose (Experimental)
  Interventions: Drug: ASP1707; Drug: Placebo
- 2 ASP1707 higher dose (Experimental)
  Interventions: Drug: ASP1707; Drug: Placebo
- 3. ASP1707 Highest dose (Experimental)
  Interventions: Drug: ASP1707; Drug: Placebo

INTERVENTIONS:
Drug: ASP1707 — oral
Drug: Placebo — oral

SUMMARY:
Three groups of 8 Japanese males are given single ascending doses of ASP1707 or placebo to assess the safety and tolerability, and to evaluate how it is absorbed, metabolized and distributed through the body.

DETAILED DESCRIPTION:
The first group receives the lowest dose while the last group receives the highest dose. ASP1707 or matching placebo is administered as a single dose under fasted conditions.

Screening takes place from Day -22 to Day -2. Subjects are admitted to the clinic on Day -1 and remain until Day 5. An end of study visit (ESV) takes place 7-14 days after discharge.

Escalation to the next higher dose takes place after review of the safety and tolerability data from the previous dose.

Safety assessments are performed throughout the study. Plasma and urine samples are collected for pharmacokinetics (PK) analysis. Serum samples are collected for pharmacodynamic (PD) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Born in Japan
* Both parents are of Japanese descent
* Time residing outside Japan does not exceed 5 years
* Maintains Japanese life style including diet
* Male subject must be non-fertile, i.e. surgically sterilized or must practice an effective contraceptive method

Exclusion Criteria:

* Subjects with out-of-range T levels in serum at screening
* Subjects with any history of cancer

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured by Adverse events (AE) | Day -2 to ESV (up to Day 19)
Safety and tolerability measured by physical examination (PE) | Day -2 to ESV (up to Day 19)
Safety and tolerability measured by vital signs (VS) | Day -2 to ESV (up to Day 19)
Safety and tolerability measured by laboratory tests | Day -2 to ESV (up to Day 19)
Safety and tolerability measured by 12 lead electrocardiogram (ECG) | Day -2 to ESV (up to Day 19)

SECONDARY OUTCOMES:
PK profile of single ascending doses of ASP1707 in plasma | Days 1 to 5
  area under the plasma concentration - time curve (AUC) extrapolated to time = infinity (AUCinf), AUC from time of dosing until last measurable concentration (AUClast), time to reach quantifiable concentrations (tlag), maximum concentration (Cmax), time to attain Cmax (tmax), terminal elimination half-life (t1/2), apparent volume of distribution (Vz/F), apparent clearance (CL/F)
PK profile of single ascending doses of ASP1707 in urine | Days 1 to 5
  amount excreted unchanged into urine (Ae) from time of dosing until last measurable concentration (Aelast), Ae extrapolated to time = infinity (Aeinf), Ae from time of dosing until last measurable concentration as percentage of total dose (Aelast%), Ae extrapolated to time = infinity as percentage of total dose (Aeinf%), renal clearance (CLR)
Pharmacodynamics of Testosterone (T) | Day -1 to ESV
  measured by minimum concentration (Cmin), time to attain Cmin (tmin), maximal %Reduction T only: number and percentage of subjects with T castration level (= T < 500 pg/mL) after single dose, time of onset and offset of T < 500 pg/mL after single dose, duration of T <500 pg/mL after single dose
Pharmacodynamics of Luteinizing Hormone (LH) | Day -1 to ESV
  measured by minimum concentration (Cmin), time to attain Cmin (tmin), maximal %Reduction T only: number and percentage of subjects with T castration level (= T < 500 pg/mL) after single dose, time of onset and offset of T < 500 pg/mL after single dose, duration of T <500 pg/mL after single dose
Pharmacodynamics of Follicle-Stimulating Hormone (FSH) levels | Day -1 to ESV
  measured by minimum concentration (Cmin), time to attain Cmin (tmin), maximal %Reduction T only: number and percentage of subjects with T castration level (= T < 500 pg/mL) after single dose, time of onset and offset of T < 500 pg/mL after single dose, duration of T <500 pg/mL after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Parexel Early Phase, Harrow, United Kingdom